CLINICAL TRIAL: NCT02291094
Title: Effect of Intravenous Infusion of Lidocaine and Remifentanil Perioperatively in Patients Undergoing Mastectomy: a Prospective, Randomized, Double-blind Study
Brief Title: Effect of Intravenous Infusion of Lidocaine and Remifentanil Perioperatively in Patients Undergoing Mastectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, MD, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Lido01
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Pain
Keywords: Intravenous lidocaine; Mastectomy; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Lidocaine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine group (Active Comparator): Patients in lidocaine group received an intravenous bolus injection of 2 mg/kg lidocaine followed by a continuous lidocaine infusion of 3 mg/kg/hr.
  Interventions: Drug: Lidocaine
- Remifentanil group (Active Comparator): Patients in remifentanil group received an intravenous bolus injection of 2 mg/kg lidocaine followed by a continuous remifentanil infusion of 0,1 mcg/kg/min.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Lidocaine — Patients in intravenous lidocaine group received an intravenous bolus injection of 2 mg/kg lidocaine followed by a continuous lidocaine infusion of 3 mg/kg/hr.
  Arms: Lidocaine group
Drug: Remifentanil — Patients in remifentanil group received an intravenous bolus injection of 2 mg/kg lidocaine followed by a continuous remifentanil infusion of 0,1 mcg/kg/min.
  Arms: Remifentanil group

SUMMARY:
This study aims to compare quality of perioperative analgesia of lidocaine and remifentanil intravenously in surgical interventions for the treatment of breast cancer.

DETAILED DESCRIPTION:
The opioid analgesics are commonly used in clinical practice for pain management in the perioperative period. However, many side effects are associated with its use, such as respiratory depression, nausea, vomiting, drowsiness, itching, urinary retention, constipation, hyperalgesia and impaired immune function. Therefore, alternative techniques and drugs have been used to replace their use. One is the intravenous infusion of lidocaine, a local anesthetic widely used in anesthetic practice. Studies show that the use of lidocaine during surgery significantly decreased postoperative pain. The mechanisms of analgesia this local anesthetic in surgical trauma may be blocking neuronal transmission in the lesion site alleviating neurogenic response, and anti-inflammatory systemic intrinsic activity. Intraoperative lidocaine promotes, besides analgesia, decreased consumption of both inhalational anesthetic and opioids; faster return of bowel movements; decreasing the production of interleukins and reduction of airway reactivity. This anesthetic also has significant anti-inflammatory properties, reduces cytokine release both in vitro and in vivo by inhibiting neutrophil activation. Besides there are few studies with use of intravenous lidocaine during the perioperative period, the intravenous injection of local anesthetic still arouses oddity among professionals; therefore, the investigators interest in the subject.

The patients underwent a prospective, randomized, double blind, in which the examiners responsible for intra and post operative will not know which group they were randomly allocated: Lidocaine group (n = 30) 3 mg / kg / h or Remifentanil group (n = 30) 0.1 mcg / kg / min.

In the clinical record, the following information will be emphasized: Blood pressure and heart rate intraoperative, perioperative side effects, quantify pain by Visual Analogue Scale (VAS) (ranging from 0 to 10 cm, zero being found when the patient is no pain and ten, with maximum or unbearable pain), Verbal Rating Scale (VRS), consisting of a list of phrases (no pain, mild pain, moderate pain, intense pain, maximum pain) and qualification of pain assessed by the amount of analgesics required postoperatively and the time to request them.

The results were analyzed statistically with the XLSTAT for Excel program using parametric and nonparametric tests, depending on the nature of the variables studied. Measures of central tendency (means) and dispersion (standard deviation) were used. The level of significance was set at < 0.05. The following tests were used: Mann-Whitney test for age, duration of anesthesia and surgery, time to first analgesic supplementation, total amount of analgesics, pain intensity; Student t-test for weight and height.

ELIGIBILITY:
Inclusion Criteria:

* Female patients scheduled for elective surgery performed mastectomy;
* Physical Status P1 and P2 of the American Society of Anesthesiology (ASA);

Exclusion Criteria:

* Patients with less than 18 years and above 75 years of age;
* Patients who are allergic to morphine and / or lidocaine;
* Patients with chronic pain;
* Patients with severe hepatic disease;
* Patients with severe renal disease;
* Patients with neurological disorders;
* Patients included in other clinical currently or within the past three months under general anesthesia studies;
* Patients who refuse to participate in the study;
* Any other condition that in the opinion of the investigator, may pose a risk to the patient or interfere with the study objectives;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of post-operative pain | Within the first 24 hours after surgery
  Quantify pain by Visual Analogue Scale (VAS, ranging from 0 to 10 cm, zero being found when the patient is no pain and ten, with maximum or unbearable pain), Verbal Rating Scale (VRS), consisting of a list of phrases (no pain, mild pain, moderate pain, intense pain, maximum pain) and qualification of pain assessed by the amount of analgesics required postoperatively and the time to request them.

SECONDARY OUTCOMES:
Evaluation of perioperative side effects | Within the first 24 hours after surgery
  Blood pressure, heart rate intraoperative, perioperative side effects

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonca, MD, Principal Investigator — Hospital de Base do Distrito Federal, Brazil

REFERENCES:
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107